CLINICAL TRIAL: NCT00167076
Title: Clinical Applications and Evaluations of A Portable In-Shoe Plantar Pressure Monitoring and Biofeedback Gait System for Ambulation Training in Stroke Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 56m2
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Stroke
Keywords: Stroke; Foot pressure; Walking speed; Gait
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purposes of this paper were to determine whether walking speed affected gait parameters and force impulse in patients with stroke or not, and if the changes varied in various foot regions.

DETAILED DESCRIPTION:
Stroke patients often suffer from persistent physical, psychological, and motor dysfunction, which severely affect their independence in daily life. Therefore, restoration of independent ambulatory ability is one of the most important goals in stroke rehabilitation. To achieve such a goal, ambulation aids are important and necessary devices to assist their ambulatory ability or ambulation training. Whereas the use of ambulation assistive devices promotes early mobility and facilitates early restoration of function for these patients, improper or prolonged use of these devices may inevitably cause negative training effects, such as patients may become over-dependent upon the assistance offered by these devices. The formation of such dependence would hinder the progress of stroke patients to achieve the ultimate goal of independent walking without any assistive devices. To assess the influences of using ambulation assistive devices, it is therefore imperative that clinicians closely and subjectively evaluate the gait pattern and force production pattern of patients when they walk with ambulation aids. In addition, ambulation assistive devices equipped with device pressure feedback function can be used not only to assist in ambulating but also to monitor patient's level of dependence on devices. The device pressure feedback information can be used to train patients to gradually reduce their dependence on devices. To date, due to the limitations of conventional laboratory methods of gait analysis, the "multi-footed" gait patterns presented by stroke patients, when they are walking with ambulation aids, have not yet been studied with biomechanical analysis. Moreover, whether the use of ambulation assistive devices equipped with feedback function can effectively improve stroke patients' gait patterns or their ability to achieve independent walking remains unknown. Answers to both questions would provide important knowledge for clinicians to base upon in evaluating weight bearing symmetry between the two lower extremities in stroke patients and the training effects of using ambulation aids for these patients.

ELIGIBILITY:
Inclusion Criteria:

* between 40 and 75 years old
* stroke confirmed by ICD-10-CM (including I60, I61, I62, I63, I67, and I63.9)
* first stroke with single side hemiplegia and received acute treatment at NTUH
* being willing to sign an informed consent approved by the Human Subjects Committee of the National Taiwan University Hospital
* able to ambulate independently and continuously for 10 meters with regular cane

Excursion criteria:

* having unstable vital sign, unconsciousness, or obvious cognitive, perception, and language impairment, and couldn't communicate with the experimenters
* having other neurological diseases, or moderate to severe neuromuscular or musculoskeletal or cardiovascular disorders, or disorders from systematic diseases other than stroke

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1999-08; Study Completion 2002-07

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Fang Tang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- School and Graduate Institute of Physical Therapy College of Medicine, National Taiwan University, Taipei, Taiwan